CLINICAL TRIAL: NCT04134845
Title: A Randomized Controlled Trial of RyR2 Inhibition With Dantrolene and Susceptibility to Ventricular Arrhythmias in Patients With Structural Heart Disease.
Brief Title: A Clinical Trial Utilizing Dantrolene in Patients With Ventricular Arrhythmias.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, William Stevenson, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190797
Record Dates: First submitted 2019-10-10; First posted 2019-10-22 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricul Tachycardia ablation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Dantrolene

STUDY DESIGN:
Intervention Model Description: 84 participants will be randomly assigned in a 2:1 ratio to treatment (dantrolene) or control (placebo). A computer-generated randomization list will be prepared by the study statistician using the stratified permuted block randomization, where block size varies randomly from 4 or 6 to ensure overall balance across treatment arms. Randomization will be stratified by 1) documented CAD with prior infarct, 2) amiodarone use within the past 21 days defined as chronic oral use or >5 grams cumulative, 3) LVEF <35%. Enrollment will be evenly distributed across the two study arms by the stratification factors
Who Masked: Participant, Investigator
Masking Description: The study statistician will generate the allocation schedule but will remain blinded to the treatment assignment as well as the study staff physician's. The research clinician will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dantrolene/Ryanodex (Experimental): Dantrolene/Ryanodex; intravenous administration of dantrolene; 1 mg/ kg IV over 3 minute, one time dose
  Interventions: Drug: Dantrolene/Ryanodex
- Placebo (Placebo Comparator): controlled placebo of saline administered Intravenous; 1 mg/kg IV over 3 minutes, one time dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dantrolene/Ryanodex — muscle relaxant
  Other Names: Dantrium, Ryanodex
  Arms: Dantrolene/Ryanodex
Drug: Placebo — Controlled placebo of saline administered Intravenous; 1 mg/kg IV over 3 minutes, one time dose
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled trial of Dantrolene (N= 84 participants) to demonstrate the feasibility of using intravenous (IV) dantrolene to study the effect of RyR2 inhibition on cardiac electrophysiology, hemodynamics, and ventricular arrhythmia inducibility in patients with structural heart disease referred for Ventricular Tachycardia (VT) ablation. The investigators will also explore the pharmacokinetic/pharmacodynamic relationship of IV dantrolene and its short-term effect on specific cardiac electrophysiologic and hemodynamic parameters.

DETAILED DESCRIPTION:
The hypothesis to be tested is that RyR2 hyperactivity in patients with structural heart disease drives proarrhythmic changes in refractoriness and conduction, and decreases cardiac contractility, which promotes Ventricular Tachycardia/Ventricular Fibrillation (VT/VF). Dantrolene, a currently available drug that inhibits RyR2, but has no Sodium (Na) or potassium (K) channel activity, will be used as a tool to study RyR2 modulation. The investigators propose a randomized controlled trial of dantrolene versus placebo in patients with structural heart disease referred for VT ablation to evaluate electrophysiologic, hemodynamic, and arrhythmia prevention endpoints. Dantrolene's inhibition of RyR1 will also be studied to define its effect on muscle and respiratory strength in this clinical population, which will be important if dantrolene is to be considered for repurposing as an antiarrhythmic drug.

The two aims are:

Aim 1: To conduct a randomized, placebo-controlled trial of dantrolene to study the effect of RyR inhibition on cardiac electrophysiology, hemodynamics, arrhythmia inducibility, muscle strength, and respiratory mechanics in patients with structural heart disease referred for Ventricular Tachycardia (VT) ablation.

Aim 2: To explore the pharmacokinetic/pharmacodynamic relationship of IV dantrolene and its short-term effect on cardiac electrophysiology, hemodynamics, and muscle and respiratory strength.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Able to give written informed consent
* Referred for catheter-based VT ablation
* Structural heart disease (cardiomyopathy or RV/LV scar)
* Permanent pacemaker or implantable cardioverter defibrillator

Exclusion Criteria:

* Mechanical ventricular support (e.g. LVAD, ECMO)
* NYHA class IV heart failure
* LVEF < 20%
* Morbid obesity (BMI > 40 kg/m2)
* Severe renal insufficiency (GFR<30 mL/min)
* Chronic liver disease (Child Pugh class A-C)
* Current use of calcium channel blockers
* Neuromuscular disorder (e.g. muscular dystrophy)
* Chronic obstructive pulmonary disease or restrictive lung disease requiring oxygen
* Therapy or history of intubation
* Pregnant or nursing
* History of dysphagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Stevenson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Harasis MA, Yoneda ZT, Varghese B, Grauherr D, Crawford DM, Schmeckpeper J, Williams HL, Ye F, Sun L, Tandri H, Richardson T, Kanagasundram A, Davogustto G, Roden D, Mantinan M, Pretorius M, Billings FT, Siegrist K, Akers WS, Stevenson WG, Knollmann BC, Shoemaker MB. Ryanodine Receptor Inhibition with Dantrolene Prevents Ventricular Tachycardia Induction in Patients with Structural Heart Disease - A Randomized Controlled Trial. medRxiv [Preprint]. 2025 Aug 19:2025.08.17.25333868. doi: 10.1101/2025.08.17.25333868. PMID 40894163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A member of the study team identified eligible subjects. Eligible subjects were identified if they were scheduled for a Ventricular Tachycardia (VT) ablation or a Premature Ventricular Contraction (PVC) ablation. The study coordinator then requested permission to contact them about research. If the patient agreed, a member of the study team would approach the patient in person in the Arrhythmia Clinic, Vanderbilt University Hospital, or by phone before ablation.
Pre-assignment Details: Sixty-eight subjects were enrolled. Fifty-one completed the protocol. 17 participants didn't receive either the drug or the placebo and were withdrawn. Nine due to a prolonged procedure, one developed hypotension, two had tachycardia, one had pulmonary concerns from anesthesia, one participant's eGFR was low, one had a drop in venous oxygen during procedure, one had safety concerns due to several cardioversion's during the procedure and one had a drop in ejection fraction.
Period: Overall Study
Arm/Group | Dantrolene/Ryanodex | Placebo
Started | 41 | 27
Completed | 29 | 22
Not Completed | 12 | 5
Not completed — withdrawl by PI | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dantrolene/Ryanodex | Placebo | Total
Number analyzed (Participants) | 29 | 22 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 19 | 15 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.2 [61.2 to 73.2] | 67.0 [62.8 to 73.6] | 67.8 [61.7 to 73.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 28 | 21 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 25 | 20 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: 17 participants did not receive either the drug or the placebo and were withdrawn from the RCT. Nine due to a prolonged procedure, one developed hypotension, two had tachycardia, one had pulmonary concerns from anesthesia, one participant's eGFR was low, one had a drop in venous oxygen during procedure, one had safety concerns due to several cardioversion's during the procedure and one had a drop in ejection fraction.
  participants
    United States | 29 | 22 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inducible Sustained Ventricular Tachycardia/ Ventricular Fibrillation (VT/VF) Utilizing Standardized Stimulation Protocol.
Description: Post drug ventricular stimulation with Right Ventricle (RV) ventricular catheter in the Right Ventricle( RV) apex with increasing extra stimuli with planned decrement stimuli by 10 milliseconds (ms) to effective refractory period (ERP). Outcome is measured as Ventricular inducibility yes/no.
Time Frame: 10 minutes post drug infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Dantrolene/Ryanodex | Placebo
Number analyzed (Participants) | 29 | 22
Participants | 4 | 9

2. Secondary Outcome: Stage of Inducibility of Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) by Standardized Ventricular Stimulation Protocol Pre and Post Drug/Placebo.
Description: A standardized induction protocol is performed using programmed ventricular stimulation from the Right Ventricular apex which was done pre-drug/placebo and post drug/placebo. The induction is single, double or triple extra beats of stimulation.
Time Frame: 10 minutes post drug infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Dantrolene/Ryanodex | Placebo
Number analyzed (Participants) | 29 | 22
Participants
  Single extra beats/ pre drug/placebo | 0 | 1
  Single extra beats/post drug/placebo | 0 | 1
  Double extra beats/pre drug/placebo | 2 | 4
  Double extra beats/post drug/placebo | 1 | 3
  Triple extra beats/pre drug/placebo | 10 | 5
  Triple extra beats/post drug/placebo | 3 | 5

3. Other Pre Specified Outcome: Serial Heart Rate Measurements
Description: Heart rate measurement performed by standard heart rate monitors in the Electrophysiology lab.
Time Frame: pre drug infusion, 1 minute, 5 minute, 10 minute and 20 minutes post infusion
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Participants With a Change of Blood Pressure
Description: Change in serial blood pressure at specified time points.
Time Frame: 1 minute, 5 minute,10 minute, 15 minute and 20 minutes post infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Dantrolene/Ryanodex | Placebo
Number analyzed (Participants) | 29 | 22
Participants
  1 minute | 0 | 0
  5 minutes | 0 | 0
  10 minutes | 0 | 0
  15 minutes | 0 | 0
  20 minutes | 0 | 0

5. Other Pre Specified Outcome: Serial Arterial O2 Sats
Description: Hemodynamic monitoring for O2 sats will be performed during ablation with an arterial line and pulmonary artery (PA) catheter (aka. Swann-Ganz Catheter).
Time Frame: pre drug, post drug 1 minute, 5 minute, 10 minute and 20 minutes
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Serial Mixed Venous O2 Sats- Measured From PA Catheter
Description: Hemodynamic monitoring for mixed venous O2 sats will be performed during ablation with an arterial line and pulmonary artery (PA) catheter (aka. Swann-Ganz Catheter).
Time Frame: pre drug infusion, 1 minute , 5 minute, 10 minute and 20 minutes post drug infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Serial PA Measurements
Description: PA- mmHg; Hemodynamic monitoring for PA will be performed during ablation with an arterial line and pulmonary artery (PA) catheter (aka. Swann-Ganz Catheter).
Time Frame: pre drug infusion , 1 minute, 5 minute, 10 minute and 20 minutes post drug infusion
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Serial Pulmonary Cap. Wedge Pressure Measurements
Description: Measuring the Pulmonary Capillary Wedge pressure by the hemodynamic pulmonary cathether
Time Frame: pre drug infusion, 1 minute, 5 minute, 10 minute and 20 minutes post drug infusion
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Per the Pharmacokinetics Measurements That Will be Collected and Measured Offline-drug Half Life
Description: The pharmacokinetic measurement of the time it takes for the concentration of the drug in the body to decrease by half.
Time Frame: post drug infusion at 5 minutes,10 minutes,15 minutes, 20 minutes, 1-4 hours, 6-12 hours,16-24 hours and optional 28-36 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Maximum Observed Plasma Concentration
Description: A pharmacokinetic measure to determine the highest concentration of the drug.
Time Frame: Post drug infusion at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 1-4 hours, 6-12 hours,16-24 hours and optional 28-36 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration
Description: Tmax (h) Time to maximum concentration by plasma concentration.
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Area Under the Concentration-time Curve From Zero to Infinity
Description: A measurement of pharmacokinetics which is the area under the curve measured as a function of time.
Time Frame: as for outcome 10
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Ventricular Effective Refractory Period Pre/Post Dantrolene
Description: Ventricular effective refractory period measured via electrophysiology catheter.
Time Frame: pre-drug infusion, post drug infusion at 5 minutes, 10 minutes,15 minutes and 20 minute post-drug
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Oxygen Saturation
Description: Oxygen saturation measured by pulse oximeter, %
Time Frame: pre-procedure, during procedure
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Respiratory Rate
Description: Rate of respiration, respiration per minute
Time Frame: pre-procedure, during procedure
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Minute Ventilation
Description: Ventilator measured L/min of ventilation
Time Frame: during procedure
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Tidal Volume
Description: Volume of ventilated air, measured as L/breath
Time Frame: during procedure
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Arterial Blood Gas - pH
Description: Blood gas, obtained from arterial blood supply, pH measurement
Time Frame: pre-procedure, during procedure, two hours post procedure
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Arterial Blood Gas - pO2
Description: Blood gas, obtained from arterial blood supply, mmHg of O2 concentration
Time Frame: Pre-procedure, during procedure, two hours post procedure
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Arterial Blood Gas - pCO2
Description: Blood gas, obtained from arterial blood supply, mmHg of CO2 concentration
Time Frame: pre-procedure, during procedure, two hours post procedure
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Arterial Blood Gas - Base Excess
Description: Blood gas, obtained from arterial blood supply, mmHg of CO2 concentration
Time Frame: pre-procedure, during procedure, two hours post procedure
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Muscle Strength
Description: Handgrip strength using a dynamometer; measured in pounds of force
Time Frame: pre-procedure, two hours post procedure
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Neuromuscular Twitch Height
Description: Twitch amplitude; measured as a % of the baseline calibration twitch amplitude (unitless, % change)
Time Frame: During procedure, post drug infusion at 0, 5, 10, 15, 20 minutes
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Respiratory Support
Description: Bag/mask ventilation, CPAP, BiPAP, LMA, or tracheal intubation
Time Frame: pre-procedure, during procedure, and two hours post procedure
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Negative Inspiratory Force
Description: Measured by bedside breathing test.
Time Frame: pre-procedure and two hours post procedure
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Neuromuscular Train of Four
Description: Train of four stimulation test measured as a % of the fourth stimulation compared to the first (unitless, % change)
Time Frame: pre-procedure, during procedure, post drug infusion at 0, 5, 10, 15, 20 minutes, and continuous
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Blood Chemistry
Description: Arterial blood concentrations of sodium, chloride, potassium, ionized calcium, bicarbonate, glucose, and lactate measured in SI ) international system of units.
Time Frame: pre-procedure, during procedure, two hours post procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours post ablation
Arm/Group | Dantrolene/Ryanodex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/22
Other Adverse Events (participants affected / at risk) | 5/29 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dantrolene/Ryanodex (N=29) | Placebo (N=22)
Intensive Care Unit (Cardiac disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04134845/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04134845/ICF_002.pdf